CLINICAL TRIAL: NCT01356394
Title: Weight Loss Improves Renal Hemodynamics in Patients With Metabolic Syndrome
Brief Title: Weight Loss Improves Renal Hemodynamics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nucleus of Education Interdisciplinary Research and Treatment in Nephrology (Other)
Collaborators: Federal University of Juiz de Fora (Other)
Responsible Party: Ezequiel, DGA, professor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 273/2006
Record Dates: First submitted 2011-05-11; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Metabolic Syndrome; Chronic Kidney Disease
Keywords: Obesity; Metabolic Syndrome; Microalbuminuria; Chronic Kidney Disease
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Renal Insufficiency, Chronic | interventions — Diet Therapy; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: dietary intervention — 12-week calorie-restricted diet consisting of 50% carbohydrate, 20-25% protein, and 25-30% fat
  Other Names: calorie-restricted diet

SUMMARY:
Metabolic syndrome (MS) is a clustering of risk factors for cardiovascular disease (CVD) such as hypertension, hypertriglyceridemia, low HDL-cholesterol levels, disorders of glucose metabolism, and insulin resistance. A number of associated conditions are included in the MS spectrum such as abdominal obesity, systemic inflammatory activation, endothelial dysfunction, non-alcoholic fatty liver disease, hyperuricemia, polycystic ovarian syndrome, and microalbuminuria. As a consequence, the diagnosis of MS identifies patients who are at increased risk for type 2 diabetes mellitus and CVD. In the last few years, the potential for MS to trigger renal damage and accelerate the progression of pre-existing nephropathy has become a focus of research. Some studies have suggested that MS can influence the development of CKD, although the underlying mechanisms are not well understood. In this study, the investigators hypothesized that modifying a key component of the MS, namely obesity, could attenuate renal damage. The investigators examined the impact of weight loss on creatinine clearance and urinary albumin excretion in non-diabetic obese patients with MS.

DETAILED DESCRIPTION:
Non-diabetic patients with MS were recruited from an outpatient clinic at the Division of Nephrology of the Federal University of Juiz de Fora, Brazil. MS was defined according to the criteria of the National Cholesterol Education Program Adult Treatment Panel III (NCEP-ATPIII). The study was divided into two phases: phase 1 (baseline) and phase 2 (intervention). At the first study visit, a full medical history was taken and a clinical examination was performed. Blood samples were taken to determine plasma glucose levels, both after fasting and 2 h after a 75-g oral glucose overload (oral glucose tolerance test; OGTT), as well as levels of plasma insulin, creatinine, total cholesterol, HDL-cholesterol, triglycerides, and uric acid. At visit 2, the preliminary results were evaluated and urine samples were collected in duplicate for measurement of microalbuminuria. Creatinine clearance was estimated using the Cockcroft-Gault formula, corrected for body surface area. The subjects were kept free of any medication (statins, antihypertensive, and anti-inflammatory drugs) over the entire study period. The only medications allowed during the study were analgesics such as dipyrone and hioscin. At visit 3, each patient was evaluated by a registered dietitian with expertise in medical nutrition therapy with the aim of achieving a weight loss of at least 5% from baseline. Patients were commenced on a 12-week calorie-restricted diet consisting of 50% carbohydrate, 20-25% protein, and 25-30% fat. The patients were evaluated by the dietitian every 2 weeks. At the final visit all laboratory tests were repeated. At the end of phase 2, patients were divided into two groups: responders, who had achieved at least a 5% reduction in body weight and non-responders, who had not achieved the target weight reduction.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age: 20 to 65 years old
* Metabolic syndrome according to the criteria of the National Cholesterol Education Program Adult Treatment Panel III

Exclusion Criteria:

* fasting plasma glucose > 126 mg/dL or a history of diabetes mellitus
* hypertension stage 2 or 3
* glomerulonephritis
* CKD stages 3, 4, or 5
* severe heart or lung disease
* pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Renal Hemodynamics | 12 weeks
  Hemodynamics renal parameters, namely, creatinine clearance and urinary albumin excretion were measured before and after twelve weeks on a calorie restricted diet.

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio B de Paula, PhD, Principal Investigator — professor
Locations (1):
- NIEPEN, Juiz de Fora, Minas Gerais, Brazil